CLINICAL TRIAL: NCT00591734
Title: A Phase II Trial of RAD001 Plus Bevacizumab in the Treatment of Patients With Metastatic Melanoma
Brief Title: RAD001 Plus Bevacizumab in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MEL 16
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; Everolimus; RAD001; Bevacizumab
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All patients received bevacizumab 15 mg/kg, administered by intravenous (IV) infusion on day 1 of each 21 day course. In addition, patients received everolimus 10 mg orally on a daily basis.
  Interventions: Drug: Bevacizumab; Drug: Everolimus

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg of bevacizumab intravenously (IV) once every 3 weeks.
  Other Names: Avastin
Drug: Everolimus — 10 mg by mouth daily
  Other Names: Afinitor; RAD001

SUMMARY:
This is a non-randomized, open label Phase II study comparing bevacizumab and everolimus in the treatment of metastatic melanoma.

DETAILED DESCRIPTION:
All patients will begin treatment with the same doses of RAD001 and bevacizumab. Patients will receive 6 weeks of treatment, followed by re evaluation. Patients with objective response or stable disease will continue treatment until disease progression.

During the study, all patients will receive 10 mg of RAD001 orally daily and 15 mg/kg of bevacizumab intravenously (IV) once every 3 weeks.

Fifty-five patients will be enrolled in this multi-centered study

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed melanoma.
2. Unresectable stage IV disease, or recurrent disease with metastases.
3. Measurable disease (by Response Evaluation Criteria in Solid Tumors [RECIST]) or measurable skin lesions.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
5. Life expectancy >=12 weeks.
6. Patients are allowed 0-2 prior treatment regimens containing chemotherapy and/or immunotherapy (interferon, interleukin 2).
7. Women of childbearing potential must have a negative serum pregnancy test with 7 days before beginning treatment.
8. Absolute neutrophil count (ANC) >=1500/µL, and platelets >=100,000/µL.
9. Serum creatinine <=2.0 mg/dL.
10. Serum bilirubin <=1.5 mg/dL institutional upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 × ULN or <5 × ULN in patients with documented liver metastases.

Exclusion Criteria:

1. Previous treatment with bevacizumab or other anti-angiogenesis agents.
2. Previous treatment with mTOR inhibitors.
3. Drugs or substances known to be inhibitors or inducers of the isoenzyme CYP3A are not allowed.
4. Treatment with investigational agents within 4 weeks of study entry.
5. Treatment with more than two previous chemotherapy regimens.
6. Immunization with attenuated live vaccines within one week of study or anytime during study treatment period.
7. Female patients who are pregnant or breastfeeding.
8. Central nervous system (CNS) involvement by metastatic melanoma.
9. CNS disease (e.g., seizures not controlled with standard medical therapy, history of stroke).
10. Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

    * Severely impaired lung function.
    * Uncontrolled diabetes as defined by fasting serum glucose >1.5 ULN,
    * Any acute or chronic uncontrolled infection/disorder.
    * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardize by the treatment with the study therapy.
    * Any acute or chronic uncontrolled infection/disorder.
    * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardize by the treatment with the study therapy.
    * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
11. Acute myocardial infarction (MI) with the previous 6 months.
12. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, unstable angina, New York Heart Association [NYHA] Class II or greater congestive heart failure [CHF], serious cardiac arrhythmia requiring medication), or >= grade 2 vascular disease.
13. Clinical history of hemoptysis or hematemesis.
14. Clinical evidence or history of a bleeding diathesis or coagulopathy.
15. Major surgical procedures, fine-needle aspirations, or core biopsies with 7 days of starting treatment.
16. Patients with PEG tubes or G-tubes.
17. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
18. Proteinuria at screening as demonstrated by either

    1. Urine protein:creatinine (UPC) ratio >= 1.0 at screening OR
    2. Urine dipstick for proteinuria >= 2+ (patients discovered to have >=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate <= 1g of protein in 24 hours to be eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (15):
- United States (15):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - Consultants in Medical Oncology and Hematology, Drexel Hill, Pennsylvania
  - Chattanooga Oncology & Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Result] Hainsworth JD, Infante JR, Spigel DR, Peyton JD, Thompson DS, Lane CM, Clark BL, Rubin MS, Trent DF, Burris HA 3rd. Bevacizumab and everolimus in the treatment of patients with metastatic melanoma: a phase 2 trial of the Sarah Cannon Oncology Research Consortium. Cancer. 2010 Sep 1;116(17):4122-9. doi: 10.1002/cncr.25320. PMID 20564157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 57
Completed | 4
Not Completed | 53
Not completed — Lack of Efficacy | 35
Not completed — Adverse Event | 5
Not completed — Physician Decision | 5
Not completed — Intercurrent Illness | 8

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 57
Age, Continuous [Median (Full Range); unit: years] | 70 [36 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Length of time, in months, that patients were alive from their first date of protocol treatment until worsening of their disease
Time Frame: 13 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intervention
Number analyzed (Participants) | 57
months | 4 [2.8 to 5.3]

2. Secondary Outcome: Overall Survival Rate
Description: Overall Survival is defined as the length of time, in months, that patients were alive from their first date of protocol treatment until death. For patients who were alive at the time of calculation, follow-up time was censored at date of last contact. The percentage of patients who were alive at 1 year is reported here. This was estimated using the Kaplan Meier method.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 57
percentage of participants | 43

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of patients who experience an objective benefit from treatment (CR+PR). The response categories were assigned using RECIST criteria. Complete Response (CR) = Disappearance of all target lesions ; Partial Response (PR) = >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 57
Participants | 7

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 29/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=57)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest, non-fatal (Cardiac disorders) | 1 (1)
Coagulation - Other (Blood and lymphatic system disorders) | 1 (1) — Coagulopathy
Fever (General disorders) | 2 (2)
Weakness (General disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Death (General disorders) | 3 (3)
Pain - Abdomen (General disorders) | 5 (5)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
GI - Other (Gastrointestinal disorders) | 1 (1) — Zenker's diverticulum
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 3 (5)
Angioedema (Immune system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Pain - Chest (General disorders) | 2 (2)
Pain - GI (General disorders) | 1 (1)
Pain - Head (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1)
Thrombus/Thrombosis/Embolism (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=57)
Albumin (Metabolism and nutrition disorders) | 9 (20)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 7 (16)
Allergic Reaction (Immune system disorders) | 4 (10)
ALT (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 27 (78)
AST (Metabolism and nutrition disorders) | 6 (9)
Cholesterol (Metabolism and nutrition disorders) | 18 (74)
Confusion (Psychiatric disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 13 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (64)
Creatinine (Metabolism and nutrition disorders) | 5 (9)
Dehydration (Gastrointestinal disorders) | 6 (8)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 25 (60)
Dyspepsia (Gastrointestinal disorders) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (46)
Edema: Head and Neck (Blood and lymphatic system disorders) | 5 (7)
Edema - Limb (Blood and lymphatic system disorders) | 17 (51)
Fatigue (General disorders) | 38 (144)
Fever (General disorders) | 9 (10)
Hemoglobin (Blood and lymphatic system disorders) | 28 (102)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 14 (23)
Hemorrhage - Hematuria (Blood and lymphatic system disorders) | 4 (6)
Hemorrhoids (Gastrointestinal disorders) | 5 (13)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (34)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Cardiac disorders) | 15 (72)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 15 (53)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 6 (11)
Hyponatremia (Metabolism and nutrition disorders) | 7 (18)
Infection - Pneumonia (Infections and infestations) | 3 (4)
Infection - Renal/Genitourinary (Infections and infestations) | 4 (6)
Infection with Normal ANC (Infections and infestations) | 7 (16)
INR (Blood and lymphatic system disorders) | 4 (10)
Insomnia (General disorders) | 6 (21)
Leukocytes (Blood and lymphatic system disorders) | 21 (44)
Mood Alteration - Depression (Psychiatric disorders) | 4 (9)
Mucositis/Stomatitis (Gastrointestinal disorders) | 31 (81)
Nausea (Gastrointestinal disorders) | 19 (42)
Neuropathy - Sensory (Nervous system disorders) | 4 (13)
Neutrophils (Immune system disorders) | 6 (8)
Pain - Abdomen (General disorders) | 12 (23)
Pain - Back (General disorders) | 7 (10)
Pain - Chest (General disorders) | 8 (16)
Pain - Dental (General disorders) | 6 (9)
Pain - GI (General disorders) | 6 (11)
Pain - Head (General disorders) | 15 (29)
Arthralgia (General disorders) | 5 (14)
Pain - Limb (General disorders) | 15 (50)
Myalgia (General disorders) | 6 (9)
Platelets (Blood and lymphatic system disorders) | 28 (75)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Proteinuria (Metabolism and nutrition disorders) | 22 (51)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (13)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 26 (86)
Taste Alteration (Gastrointestinal disorders) | 9 (35)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 13 (18)
Weakness (General disorders) | 3 (4)
Weight Loss (Metabolism and nutrition disorders) | 10 (28)
Wound Complication (Skin and subcutaneous tissue disorders) | 3 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.